CLINICAL TRIAL: NCT03587844
Title: Optimizing Dosing of Brentuximab Vedotin for Mycosis Fungoides, Sezary Syndrome, and Lymphomatoid Papulosis
Brief Title: Dosing of Brentuximab Vedotin for Mycosis Fungoides, Sezary Syndrome Patients
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Seagen Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 18-147
Record Dates: First submitted 2018-07-03; First posted 2018-07-16 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Mycosis Fungoides; Lymphomatoid Papulosis; Sezary Syndrome
Keywords: Brentuximab Vedotin; 18-147
MeSH Terms: conditions — Mycosis Fungoides; Lymphomatoid Papulosis; Sezary Syndrome | interventions — Brentuximab Vedotin

STUDY DESIGN:
Intervention Model Description: Following identification of a promising dose after the completion of the full Cohort 1 Simon two stage design, enrollment will initiate onto cohort 2 at the dose found to be promising in cohort 1. If neither dose is found promising, cohort 2 will not start.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (3):
- not been previously treated with brentuximab vedotin. (Experimental): Patients with MF/SS who have not been previously treated with brentuximab vedotin. For MF patients: Treatment delays lasting longer than 8 weeks for toxicity will result in removal from study. As of October 2020, the Simon two stage design for Cohort 1 has restarted at the 1.2 mg/kg dose.
  Interventions: Drug: brentuximab vedotin
- treated with reduced dose brentuximab vedotin (Experimental): Patients with MF/SS who were previously treated with brentuximab vedotin. Up to 10 patients will be enrolled onto this cohort. Following identification of a promising dose after the completion of the full Cohort 1 Simon two stage design, enrollment will initiate onto cohort 2 at the dose found to be promising in cohort 1. For MF patients: Treatment delays lasting longer than 8 weeks for toxicity will result in removal from study. The 0.9mg/kg dose did not meet the primary endpoint for response, therefore 1.2 mg/kg has been chosen as the dose for Cohort 2. As of October 2020, enrollment on our exploratory Cohort 2 has opened at the 1.2 mg/kg dose.
  Interventions: Drug: brentuximab vedotin
- Patients with LyP (Experimental): Patients with LyP patients with lymphomatoid papulosis will receive brentuximab vedotin 0.9 mg/kg as an intravenous infusion over 30 minutes every three weeks. Cohort 3 will enroll patients concurrently with Cohort 1. Treatment may be held if felt to be in patient's best interest (for example: for toxicity or no active disease). Treatment can be reinitiated after discussion with MSK PI as long as the study is still open and patient has not received alternate systemic therapy.
  Interventions: Drug: brentuximab vedotin

INTERVENTIONS:
Drug: brentuximab vedotin — MF/SS Brentuximab vedotin 0.9 mg/kg 0R 1.2 mg/kg.
  Arms: not been previously treated with brentuximab vedotin.
Drug: brentuximab vedotin — LyP Brentuximab vedotin 0.9 mg/kg2
  Arms: Patients with LyP
Drug: brentuximab vedotin — MF/SS prior brentuximab vedotin-Brentuximab vedotin dose to be determined from Cohort 1
  Arms: treated with reduced dose brentuximab vedotin

SUMMARY:
The purpose of this study is to test any good and bad effects of the study drug called brentuximab vedotin at a lower dose than is FDA-approved.

ELIGIBILITY:
Inclusion Criteria:

Mycosis fungoides (MF) and Sezary Syndrome (SS)

1. Pathologically confirmed mycosis fungoides/sezary syndrome at the enrolling institution, disease stage IB (defined as patches, plaque, or papules that involve 10% of the skin surface viscera) or higher

   ° CD30 negative mycosis fungoides patients are eligible.
2. Age ≥ 18 years
3. ECOG Performance Score ≤ 2
4. For Cohort 1, patients who have not received brentuximab vedotin are eligible.
5. For Cohort 2, patients who have previously had brentuximab vedotin for MF/SS are eligible. Patients previously treated on Cohort 1 who were discontinued due to toxicity are not eligible for Cohort 2.
6. Previous systemic anti-cancer therapy must have been discontinued at least 2 weeks prior to treatment.

   ° See section 6.2 Subject Exclusion Criteria for guidelines regarding adjuvant and maintenance therapy for prior malignancy.
7. Topical or systemic steroids (equivalent to ≤ 10 mg/day of prednisone) may be considered if dose has been constant and discontinuation may lead to rebound flare in disease, adrenal insufficiency, and/or unnecessary suffering, after discussion with PI.
8. If HIV+, patient must be on stable anti-retroviral treatment for 12 weeks prior to C1D1, with CD4 count >200 within 7 days prior to C1D1.
9. Females of childbearing potential must be on acceptable form of birth control per instutional standard.

Lymphomatoid papulosis (LyP)

1. Pathologically confirmed lymphomatoid papulosis at the enrolling institution
2. Requiring systemic treatment per investigator's discretion
3. Age ≥ 18 years
4. ECOG Performance Score ≤ 2
5. Previous systemic anti-cancer therapy must have been discontinued at least 2 weeks prior to treatment.
6. Topical or systemic steroids (equivalent to ≤ 10 mg/day of prednisone) may be considered if dose has been constant and discontinuation may lead to rebound flare in disease, adrenal insufficiency, and/or unnecessary suffering.
7. If HIV+, patient must be on stable anti-retroviral treatment for 12 weeks prior to C1D1, with CD4 count >200 within 7 days prior to C1D1.
8. Females of childbearing potential must be on acceptable form of birth control per institutional standard

Exclusion Criteria:

1. Concurrent use of other systemic anti-cancer agents or treatments for mycosis fungoides/sezary syndrome, or lymphomatoid papulosis.
2. Grade 2 or greater neuropathy
3. Severe renal impairment (CrCL <30 mL/min)
4. Moderate or severe hepatic impairment (Child-Pugh B or Child-Pugh C)

   ° See Appendix E for Child Pugh Classification chart
5. Women of reproductive potential† must have a negative Serum ß human chorionic gonadotropin (ß-HCG) pregnancy test within 1 week of C1D1. They should discuss contraception with treating provider.
6. Previous use of brentuximab vedotin (for Cohort 1 ONLY)
7. Receiving systemic therapy for another primary malignancy (other than T-cell lymphoma).

   * Patients with more than one type of lymphoma may be enrolled after discussion with the MSK Principal Investigator.
   * Adjuvant or maintenance therapy to reduce the risk of recurrence of other malignancy (other than T-cell lymphoma) is permissible after discussion with the MSK Principal Investigator.
8. For Cohort 2, patients who previously progressed on the standard 1.8mg/kg dose and schedule of brentuximab vedotin are ineligible.

   * A female of reproductive potential is a sexually mature female who: has not undergone a hysterectomy or bilateral oophorectomy; or has not been naturally postmenopausal for at least 24 consecutive months (i.e. has had menses at any time in the preceding 24 consecutive months).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 58 (Estimated)
Dates: Start 2018-07-03 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
overall response | 1 year
  measure best overall response during treatment by the global response score, which incorporates the mSWAT, as well as CT scan for patients with baseline nodal/visceral involvement and flow cytometry for patients with baseline positive peripheral flow cytometry

CONTACTS AND LOCATIONS:
Overall Officials: Alison Moskowitz, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Stanford University Medical Center, Stanford, California
  - Memorial Sloan Kettering Basking Ridge, Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth, Middletown, New Jersey
  - Memorial Sloan Kettering Bergen, Montvale, New Jersey
  - Memorial Sloan Kettering Commack, Commack, New York
  - Memorial Sloan Kettering Westchester, Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau, Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/mskcc/html/44.cfm